CLINICAL TRIAL: NCT06068140
Title: Evaluation of the Effectiveness of the Complex of Carnitine Orotate and Biphenyl Dimethyl Dicarboxylate in the Adjuvant Therapy of Chronic Hepatitis D in Real Clinical Practice: a Prospective Cohort Study
Status: Withdrawn | Type: Observational
Why Stopped: Administartive issues
Sponsor: Kazakh Association of Internal Medicine Specialists (Other)
Responsible Party: Sponsor
Other Study IDs: KAIMS-02
Record Dates: First submitted 2023-09-26; First posted 2023-10-05 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2023-09

CONDITIONS: Chronic Viral Hepatitis B With Delta-Agent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Cohort: Patients taking Carnitine-Orotate Complex and Biphenyl Dimethyl Dicarboxylate
- Control cohort: Patients who do not take Carnitine-Orotate Complex and Biphenyl Dimethyl Dicarboxylate

SUMMARY:
The goal of this observational study is to evaluate the effectiveness of the carnitine-orotate complex and biphenyl dimethyl dicarboxylate in the adjuvant therapy of chronic hepatitis D in real clinical practice: a prospective cohort study

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 18 to 75 years who are citizens of the Republic of Kazakhstan;
* An established diagnosis of CGD (chronic viral hepatitis B with the delta agent);
* Patients who have contraindications to taking peg-INF-alpha2a and/or have failed treatment with peg-INF-alpha2a;
* Compensated liver disease ≤ CPT A (6 points);
* Patients without severe concomitant diseases;
* Patients who do not receive other adjuvant therapy (metabolic therapy drugs, essential phospholipids, ursodeoxycholic acid, glycyrrhizic acid, ademetionine and others);
* Patients who voluntarily signed the informed consent form.

Exclusion Criteria:

* Patients taking COC for more than 4 weeks before inclusion in the study;
* Patients with contraindications to the COC;
* Decompensated liver disease severity class > CPT A6;
* Patients taking peg-IFN-alpha 2a;
* Alcohol abuse according to the AUDIT-c questionnaire;
* Pregnancy and lactation;
* Patients with coinfection with HIV, HCV;
* GFR ≤ 15 ml/min/1.73 m2;
* Exclude patients with significant biochemical activity (ALT, AST more than 10 ULN) and total bilirubin more than 2 norms;
* Patients with other causes of liver damage;
* Drug addict people;
* Malignant formations of the liver and other organs (in history and currently) or a clinically significant increase in alpha-fetoprotein more than 5 times or more;
* Patient takes part in an interventional clinical trial.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Persons aged ≥18 to 75 years inclusive with a diagnosis of chronic hepatitis D who are undergoing outpatient monitoring at the place of residence.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
1. Normalization of ALT levels during adjuvant CGD therapy at 12 months among study participants taking and not taking COC and BDD | at 12 months

SECONDARY OUTCOMES:
Normalization of ALT levels during adjuvant CGD therapy at 6 months among study participants taking and not taking COCs AND BDD | at 6 months
Dynamics of the level of fibrosis during adjuvant CGD therapy at 6 and 12 months among study participants taking and not taking COCs AND BDD | at 6 and 12 months
Viral load during adjuvant CGD therapy at 6 and 12 months among study participants taking and not taking COC and BDD | at 6 and 12 months
Adherence to COC and BDD therapy against the background of adjuvant CGD therapy among study participants taking and not taking COCs and BDD | up to 12 months since enrollment
Dynamics of changes in the total score of the quality of life questionnaire | up to 12 months since enrollment
Incidence of adverse and serious unexpected adverse reactions associated with the use of COC and BDD | up to 12 months since enrollment
Satisfaction of patients with CGD with combination therapy of COCs and BDD | up to 12 months since enrollment

CONTACTS AND LOCATIONS:
Locations (7):
- Kazakhstan (7):
  - State-owned public enterprise with the right of economic management "Enbekshikazakh Interdistrict Multidisciplinary Hospital", Esik, Almaty Region
  - Karasai interdistrict multidisciplinary hospital, Kaskelen, Almaty Region
  - State-owned public enterprise with the right of economic management Regional infectious hospital of the state institution "Healthcare Department of the Almaty region", Taldykorgan, Zhetisu Region
  - LLP "InkarMed", Aktobe
  - Hepatology center on the basis of the State Public Enterprise at the RV "City Clinic No. 5", Almaty
  - Medical Center "iClinic", Astana
  - State-owned public enterprise with the right of economic management "Regional Clinical Hospital" of the Department of Public Health of the Turkestan region, Turkestan